CLINICAL TRIAL: NCT01009918
Title: Phase II Placebo-controlled Trial of Lisinopril and Coreg CR® to Reduce Cardiotoxicity in Patients With Breast Cancer Receiving (Neo)Adjuvant Chemotherapy With Trastuzumab (Herceptin®)
Brief Title: Lisinopril or Coreg CR® in Reducing Side Effects in Women With Breast Cancer Receiving Trastuzumab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SCUSF 0806; SCUSF-0806 (Other: SunCoast CCOP Research Base); 5U10CA081920-11 (NIH)
Record Dates: First submitted 2009-11-06; First posted 2009-11-09 (Estimated); Results first posted 2021-03-30 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2019-04

CONDITIONS: Breast Cancer; Cardiac Toxicity
Keywords: cardiac toxicity; HER2-positive breast cancer; recurrent breast cancer; stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; male breast cancer
MeSH Terms: conditions — Breast Neoplasms; Cardiotoxicity; Breast Neoplasms, Male | interventions — Carvedilol; Lisinopril

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm I lisinopril (Experimental): Patients receive oral lisinopril once daily.
  Interventions: Drug: lisinopril
- Arm II Coreg CR® (Experimental): Patients receive oral Coreg CR® once daily.
  Interventions: Drug: Coreg CR®
- Arm III placebo (Placebo Comparator): Patients receive oral placebo once daily.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Coreg CR® — Given orally
  Other Names: carvedilol phosphate extended-release
  Arms: Arm II Coreg CR®
Drug: lisinopril — Given orally
  Other Names: Registered Trade names: Prinivil, Tensopril, Zestril, Hipril
  Arms: Arm I lisinopril
Other: placebo — Given orally
  Arms: Arm III placebo

SUMMARY:
RATIONALE: Lisinopril or Coreg CR®, may help reduce side effects caused by trastuzumab. It is not yet known whether lisinopril or Coreg CR® are more effective than a placebo in reducing side effects caused by trastuzumab.

PURPOSE: This phase II trial is studying lisinopril and Coreg CR® to see how well they work compared with a placebo in reducing side effects in patients with HER2-positive breast cancer receiving trastuzumab.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* The primary objective of this study is to determine if administration of lisinopril or Coreg CR®, compared to placebo, will reduce the incidence of trastuzumab-induced cardiotoxicity, as measured by LVEF, in patients receiving adjuvant, or neoadjuvant,therapy for HER2 positive breast cancer.

Secondary

* To determine whether subjects randomized to active agent have fewer interruptions in trastuzumab therapy due to cardiomyopathy.
* To determine whether the treatment effect is consistent in anthracycline and nonanthracycline patient cohorts
* To compare changes in HRQL among the treatment groups during the study intervention
* To evaluate the long term effects on the prevention of cardiomyopathy and impact on HRQL for either or both study agents
* To compare the predictive value of troponin I and BNP in the identification of trastuzumab-induced cardiotoxicity

OUTLINE: This is a multicenter study. Patients are stratified according to chemotherapy comprising an anthracycline (yes vs no). Patients are randomized to 1 of 3 treatment arms.

* Arm I: Patients receive oral lisinopril once daily.
* Arm II: Patients receive oral Coreg CR® once daily.
* Arm III: Patients receive oral placebo once daily.

In all arms, study treatment begins with the first dose of trastuzumab and continues for up to 52 weeks or until the end of trastuzumab therapy.

Quality of life is assessed using the EORTC QLQ-C30 questionnaire at baseline, at 52 weeks (or at the end of trastuzumab therapy), and at 18 and 24 months (or 6 and 12 months after the completion of trastuzumab).

After completion of study treatment, patients are followed up at 3, 6, 9, and 12 months.

ELIGIBILITY:
INCLUSION CRITERIA

* Males and Females ≥ 18 years old diagnosed with HER2 positive breast cancer
* Scheduled to receive neoadjuvant or adjuvant trastuzumab (Herceptin®) therapy (anthracycline-containing regimens are permitted). Patients receiving Herceptin® with their chemotherapy are permitted for eligibility work-up. Taxanes are permitted. Trastuzumab (Herceptin®) therapy may be given with or after primary chemotherapy. Pertuzumab may be used in conjunction with trastuzumab.
* Left Ventricular Ejection Fraction (LVEF) ≥ 50% by MUGA scan or echocardiogram
* Adequate renal function for administration of trastuzumab-containing chemotherapy regimen.
* Sitting systolic blood pressure of > 90 mm Hg
* Pulse ≥ 60 beats/minute
* Not pregnant or breastfeeding
* Female patients of childbearing potential, who are sexually active, must have a negative pregnancy test before starting the study
* Both men and women must be willing to use effective contraception during the study. Teratogenicity is documented for both active study agents
* Able to swallow capsules

EXCLUSION CRITERIA:

* Patients with metastatic disease
* Prior treatment with trastuzumab or anthracyclines prior to this chemotherapy regimen
* Current treatment with angiotensin converting enzyme (ACE) inhibitors, angiotensin receptor blockers (ARBs), such as losartan, β-blockers or digoxin
* Known cardiac history: heart failure, myocardial infarction, radiation-induced cardiac dysfunction
* Known allergy to either ACE inhibitors or β-blockers
* History of bronchial asthma or related bronchospastic conditions
* Hereditary or idiopathic angioedema
* History of severe hypersensitivity reactions to drugs or other causes, i.e. bee stings
* This protocol does not exclude patients who are participating on other investigational studies. Refer to the local IRB guidelines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 468 (Actual)
Dates: Start 2010-03; Primary Completion 2017-08 (Actual); Study Completion 2018-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maya Guglin, MD, PhD, Study Chair — University of South Florida; Pamela N. Munster, MD, Study Chair — University of California, San Francisco
Locations (174):
- United States (174):
  - Todd Cancer Institute at Long Beach Memorial Medical Center, Long Beach, California
  - Olive View - UCLA Medical Center Foundation, Sylmar, California
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - St. Anthony Central Hospital, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - St. Mary - Corwin Regional Medical Center, Pueblo, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Ella Milbank Foshay Cancer Center at Jupiter Medical Center, Jupiter, Florida
  - Lakeland Regional Cancer Center at Lakeland Regional Medical Center, Lakeland, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - MBCCOP - Medical College of Georgia Cancer Center, Augusta, Georgia
  - Nancy N. and J. C. Lewis Cancer and Research Pavilion at St. Joseph's/Candler, Savannah, Georgia
  - Illinois CancerCare - Bloomington, Bloomington, Illinois
  - Illinois CancerCare - Canton, Canton, Illinois
  - Illinois CancerCare - Carthage, Carthage, Illinois
  - Resurrection Medical Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Illinois CancerCare - Eureka, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Illinois CancerCare - Havana, Havana, Illinois
  - Illinois CancerCare - Kewanee Clinic, Kewanee, Illinois
  - La Grange Memorial Hospital, La Grange, Illinois
  - Illinois CancerCare - Macomb, Macomb, Illinois
  - Illinois CancerCare - Monmouth, Monmouth, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Illinois CancerCare - Community Cancer Center, Normal, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Illinois CancerCare - Pekin, Pekin, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Illinois CancerCare - Peru, Peru, Illinois
  - Illinois CancerCare - Princeton, Princeton, Illinois
  - West Suburban Center for Cancer Care, River Forest, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - Bloomington Hospital Regional Cancer Institute, Bloomington, Indiana
  - Elkhart Clinic, LLC, Elkhart, Indiana
  - Michiana Hematology-Oncology, PC - Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - St. Francis Hospital Cancer Care Services, Indianapolis, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Michiana Hematology-Oncology, PC - South Bend, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center, Mishawaka, Indiana
  - Michiana Hematology Oncology PC - Plymouth, Plymouth, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC - La Porte, Westville, Indiana
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, Clive, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Covenant Cancer Treatment Center, Waterloo, Iowa
  - Lucille P. Markey Cancer Center at University of Kentucky, Lexington, Kentucky
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Mercy Hospital, Portland, Maine
  - Mercy Medical Center, Baltimore, Maryland
  - Alvin and Lois Lapidus Cancer Institute at Sinai Hospital, Baltimore, Maryland
  - Suburban Hospital, Bethesda, Maryland
  - Jordan Hospital Club Cancer Center, Plymouth, Massachusetts
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Bay Regional Medical Center, Bay City, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Singh and Arora Hematology Oncology, PC, Flint, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Great Lakes Cancer Institute - Lapeer Campus, Lapeer, Michigan
  - Clemens Regional Medical Center, Mount Clemens, Michigan
  - Mercy General Health Partners, Muskegon, Michigan
  - Northern Michigan Hospital, Petoskey, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Lakeside Cancer Specialists, PLLC, Saint Joseph, Michigan
  - Providence Cancer Institute at Providence Hospital - Southfield Campus, Southfield, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Willmar Cancer Center at Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology - Woodbury, Woodbury, Minnesota
  - Central Care Cancer Center, Bolivar, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Cancer Institute, Joplin, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - Mercy Hospital St. Louis, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Good Samaritan Cancer Center at Good Samaritan Hospital, Kearney, Nebraska
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Foundation Medical Partners, Nashua, New Hampshire
  - Oncology Center at St. Joseph Hospital, Nashua, New Hampshire
  - Dizzy Gillespie Cancer Institute at Englewood Hospital and Medical Center, Englewood, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - UMDNJ University Hospital, Newark, New Jersey
  - Franklin & Edith Scarpa Regional Cancer Center at South Jersey Healthcare, Vineland, New Jersey
  - Lovelace Medical Center - Downtown, Albuquerque, New Mexico
  - Presbyterian Cancer Treatment Center at Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Bassett Healthcare Regional Cancer Program at Mary Imogene Bassett Hospital, Cooperstown, New York
  - Charles R. Wood Cancer Center at Glens Falls Hospital, Glens Falls, New York
  - Nalitt Cancer Institute at Staten Island University Hospital, Staten Island, New York
  - Park Ridge Health, Henderson, North Carolina
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Aultman Cancer Center at Aultman Hospital, Canton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - United States Air Force Medical Center - Wright-Patterson, Wright-Patterson Air Force Base, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Cancer Care Associates - Norman, Norman, Oklahoma
  - Cancer Care Associates - Mercy Campus, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Geisinger Hazleton Cancer Center, Hazleton, Pennsylvania
  - Joan Karnell Cancer Center at Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Cancer Center at Phoenixville Hospital, Phoenixville, Pennsylvania
  - Guthrie Cancer Center at Guthrie Clinic Sayre, Sayre, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Keyserling Cancer Center at Beaufort Memorial Hospital, Beaufort, South Carolina
  - St. Francis Hospital, Greenville, South Carolina
  - Gibbs Cancer Center - Pelham, Greer, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Martha Jefferson Hospital Cancer Care Center, Charlottesville, Virginia
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - Mercy Regional Cancer Center, Janesville, Wisconsin
  - Gundersen Lutheran Center for Cancer and Blood, La Crosse, Wisconsin
  - D.N. Greenwald Center, Mukwonago, Wisconsin
  - Regional Cancer Center at Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Waukesha Memorial Hospital Regional Cancer Center, Waukesha, Wisconsin

REFERENCES:
- [Derived] Guglin M, Krischer J, Tamura R, Fink A, Bello-Matricaria L, McCaskill-Stevens W, Munster PN. Randomized Trial of Lisinopril Versus Carvedilol to Prevent Trastuzumab Cardiotoxicity in Patients With Breast Cancer. J Am Coll Cardiol. 2019 Jun 11;73(22):2859-2868. doi: 10.1016/j.jacc.2019.03.495. PMID 31171092

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I Lisinopril | Arm II Coreg CR® | Arm III Placebo
Started | 158 | 156 | 154
Completed | 134 | 132 | 124
Not Completed | 24 | 24 | 30

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I Lisinopril | Arm II Coreg CR® | Arm III Placebo | Total
Number analyzed (Participants) | 158 | 156 | 154 | 468
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.58 (10.91) | 51.58 (10.93) | 51.11 (10.32) | 51.09 (10.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 158 | 156 | 154 | 468
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 10 | 16 | 42
  Not Hispanic or Latino | 141 | 145 | 137 | 423
  Unknown or Not Reported | 1 | 1 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 3 | 0 | 4
  Asian | 3 | 6 | 3 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 14 | 5 | 15 | 34
  White | 137 | 137 | 130 | 404
  More than one race | 1 | 1 | 1 | 3
  Unknown or Not Reported | 2 | 4 | 4 | 10
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Population: Did not have information for 4 participants
  kg/m^2
    number analyzed (Participants) | 156 | 156 | 152 | 464
    (all) | 28.01 (6.86) | 28.26 (6.17) | 29.03 (5.92) | 28.43 (6.33)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Trastuzumab-Induced Cardiotoxicity After 52 Weeks of Treatment
Description: Reduction in incidence of trastuzumab-induced cardiotoxicity after 52 weeks of treatment as measured by preservation of Left Ventricular Ejection Fraction (LVEF). Number of Patients who experienced a cardiotoxicity.
Time Frame: 2 years
Population: Number of participants who experienced cardiotoxicity
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I Lisinopril | Arm II Coreg CR® | Arm III Placebo
Number analyzed (Participants) | 152 | 147 | 144
Participants | 45 | 43 | 46

2. Primary Outcome: Number of Participants With LVEF Decrease to <50%
Description: Number of Participants with Left Ventricular Ejection Fraction (LVEF) drop to <50%
Time Frame: 2 years
Population: LVEF drop to <50%
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I Lisinopril | Arm II Coreg CR® | Arm III Placebo
Number analyzed (Participants) | 152 | 147 | 144
Participants | 5 | 9 | 15

3. Secondary Outcome: Number of Patients With Trastuzumab Course Interruption
Description: Measure indicates the number of patients who had an interruption of trastuzumab for any reason
Time Frame: 2 years
Population: Number of patients who had an interruption of trastuzumab for any reason
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I Lisinopril | Arm II Coreg CR® | Arm III Placebo
Number analyzed (Participants) | 152 | 147 | 144
Participants | 27 | 24 | 40

4. Secondary Outcome: Quality-of-life Changes Between Baseline and 52-weeks
Description: Quality-of-life changes as assessed by North European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-C30), which measures the quality of life of cancer patients. Higher score indicates higher quality of life. Score range is 0-100. The questionnaire was administered at baseline and at 52 weeks.
Time Frame: 52 weeks
Population: Mean change from baseline to 52-week endpoint
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Arm I Lisinopril | Arm II Coreg CR® | Arm III Placebo
Number analyzed (Participants) | 128 | 129 | 111
Scores on a scale | 1 (23) | 2 (17) | 5 (21)

5. Secondary Outcome: Number of Participants With Cardiotoxicity-free Survival at 750 Days From Baseline
Description: Number of Participants with cardiotoxicity-free survival at 750 days from baseline
Time Frame: 2 years
Population: Number of Participants with cardiotoxicity-free survival at 750 days from baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I Lisinopril | Arm II Coreg CR® | Arm III Placebo
Number analyzed (Participants) | 152 | 147 | 144
Participants | 15 | 24 | 17

ADVERSE EVENTS:
Time Frame: AEs were collected for the duration of the study and 12 month follow-up period.
Description: Adverse Events were collected from patient at each study visit.
Arm/Group | Arm I Lisinopril | Arm II Coreg CR® | Arm III Placebo
All-Cause Mortality (participants affected / at risk) | 1/158 | 2/156 | 2/154
Serious Adverse Events (participants affected / at risk) | 5/158 | 4/156 | 6/154
Other Adverse Events (participants affected / at risk) | 104/158 | 89/156 | 82/154
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I Lisinopril (N=158) | Arm II Coreg CR® (N=156) | Arm III Placebo (N=154)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Nervous System Disorders - Other Specify (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — Stroke
Neutrophil Count Decreased (Investigations) | 0 (0) | 1 (1) | 2 (3)
Pericardial Effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Skin Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Spleen Disorder (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
White Blood Cell Count Decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I Lisinopril (N=158) | Arm II Coreg CR® (N=156) | Arm III Placebo (N=154)
Anemia (Blood and lymphatic system disorders) | 8 (21) | 11 (18) | 6 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (10) | 8 (8) | 6 (7)
Constipation (Gastrointestinal disorders) | 10 (15) | 13 (14) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 21 (22) | 12 (17) | 7 (7)
Diarrhea (Gastrointestinal disorders) | 49 (134) | 50 (81) | 32 (68)
Dizziness (Nervous system disorders) | 39 (60) | 30 (43) | 24 (53)
Dyspepsia (Gastrointestinal disorders) | 9 (9) | 9 (9) | 6 (8)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 31 (45) | 19 (28) | 21 (35)
Edema Limbs (General disorders) | 10 (10) | 16 (21) | 6 (6)
Fatigue (Gastrointestinal disorders) | 74 (130) | 63 (107) | 57 (126)
Headache (Nervous system disorders) | 19 (27) | 13 (26) | 13 (23)
Hot Flashes (Vascular disorders) | 6 (11) | 9 (10) | 7 (8)
Hypotension (Vascular disorders) | 24 (39) | 7 (11) | 4 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 12 (12) | 9 (9) | 5 (5)
Nausea (Gastrointestinal disorders) | 25 (36) | 22 (28) | 13 (16)
Pain (Gastrointestinal disorders) | 8 (14) | 8 (10) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-08-31): https://cdn.clinicaltrials.gov/large-docs/18/NCT01009918/Prot_SAP_000.pdf